CLINICAL TRIAL: NCT01422135
Title: A Pharmacokinetic Study of the Agile TCDS AG200-15 Following Weekly Application to Three Anatomical Sites (Abdomen, Buttock and Upper Torso) in Healthy Female Volunteers
Brief Title: Pharmacokinetic Study of AG200-15 Transdermal Patch to Three Anatomical Sites in Healthy Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agile Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ATI-CL15
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: PK and safety; Pharmacokinetic profile (PK) and safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Abdomen, Buttock, Upper Torso (Experimental): Patch was placed on abdomen, buttock then the upper torso excluding breast.
  Intervention: AG200-15 patch
  Interventions: Drug: AG200-15
- Abdomen, Upper Torso, Buttock (Experimental): Patch was placed on abdomen, upper torso excluding breast then the buttock.
  Intervention: AG200-15 patch
  Interventions: Drug: AG200-15
- Buttock, Abdomen, Upper Torso (Experimental): Patch was placed on the buttock, abdomen, then the upper torso excluding breast.
  Intervention: AG200-15 patch
  Interventions: Drug: AG200-15
- Buttock, Upper Torso, Abdomen, (Experimental): Patch was placed on the buttock, upper torso excluding breast then the abdomen
  Intervention: AG200-15 patch
  Interventions: Drug: AG200-15
- Upper Torso, Abdomen, Buttock (Experimental): Patch was placed on the upper torso excluding breast, abdomen then buttock.
  Intervention: AG200-15 patch
  Interventions: Drug: AG200-15
- Upper Torso, Buttock, Abdomen (Experimental): Patch was place on the upper torso excluding breast, buttock, then abdomen.
  Intervention: AG200-15 patch
  Interventions: Drug: AG200-15

INTERVENTIONS:
Drug: AG200-15 — A transdermal contraceptive delivery system for levonorgestrel (LNG) and ethinyl estradiol (EE). . A total of 3 patches will be worn during the study. Each patch will be worn for 1 week followed by a patch free week.
  Other Names: Transdermal contraceptive delivery system

SUMMARY:
This is a pharmacokinetics and safety study over 3 weekly applications.

DETAILED DESCRIPTION:
Pharmacokinetic study to evaluate the safety and pharmacokinetic profile of AG200-15 following application at three different anatomical sites (abdomen, buttock and upper torso).

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, ages 18-45 years
* Body mass index 18 - 32, and weight ≥ 110 lbs.
* Willing to use a non-hormonal method of contraception if of childbearing potential, Or have already undergone previous bilateral tubal ligation or hysterectomy
* Willing to refrain from use of alcohol and grapefruit juice from 48 hours prior to patch application until completion of each treatment period
* Willing to give informed consent to participate in study
* Hemoglobin within normal range.

Exclusion Criteria:

* Known or suspected pregnancy
* A cervical cytology smear of Papanicolaou (Pap) class III or greater or a Bethesda System report of low grade squamous intraepithelial lesions (SIL) or greater
* Smoking
* Hypertension (blood pressure >140 mm Hg systolic and/or >90 mm Hg diastolic)
* Diabetes Mellitus
* History of headaches with focal neurological symptoms
* Current or history of clinically significant depression in the last year
* Acute or chronic hepatocellular disease with abnormal liver function
* History of or existing venous and arterial thrombotic and thromboembolic disorder, vascular disease, cerebral vascular, or coronary artery disease
* Chronic use of any medication that might interfere with the efficacy of hormone contraceptives (including barbiturates, bosentan, carbamazepine, felbamate, griseofulvin, oxcarbazepine, phenytoin, rifampin, St. John's Wort, topiramate, and HIV protease inhibitors), OR use of these medications within the past 3 months prior to screening visit

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Garner, MD, Study Director — Agile Therapeutics
Locations (2):
- United States (2):
  - Lincoln, Nebraska
  - Neptune City, New Jersey

RESULTS

PARTICIPANT FLOW:
Groups:
- Lower Abdomen, Buttock, Upper Torso Excluding Breast: Subjects applied AG200-15 to Abdomen, Buttock, then Upper Torso excluding Breast
- Lower Abdomen, Upper Torso Excluding Breast, Buttock: Subjects applied AG200-15 to Abdomen, Upper Torso excluding Breast, then Buttock
- Buttock, Lower Abdomen, Upper Torso Excluding Breast: Subjects applied AG200-15 to Buttock, Abdomen, then Upper Torso excluding Breast
- Buttock, Upper Torso Excluding Breast, Lower Abdomen: Subjects applied AG200-15 to Buttock, Upper Torso excluding Breast, then Lower Abdomen.
- Upper Torso Excluding Breast, Lower Abdomen, Buttock: Subjects applied AG200-15 to Upper Torso excluding Breast, Lower Abdomen, then Buttock
- Upper Torso Excluding Breast, Buttock, Lower Abdomen: Subjects applied AG200-15 to Upper Torso excluding Breast, Buttock, then Lower Abdomen
Period: Overall Study
Arm/Group | Lower Abdomen, Buttock, Upper Torso Excluding Breast | Lower Abdomen, Upper Torso Excluding Breast, Buttock | Buttock, Lower Abdomen, Upper Torso Excluding Breast | Buttock, Upper Torso Excluding Breast, Lower Abdomen | Upper Torso Excluding Breast, Lower Abdomen, Buttock | Upper Torso Excluding Breast, Buttock, Lower Abdomen
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- AG200-15: Subjects will be randomly assigned to one of six treatment (site of application) sequences. Each sequence will include three patch application sites: abdomen, buttock, or upper torso excluding breasts.
  AG200-15: A transdermal contraceptive delivery system for levonorgestrel (LNG) and ethinyl estradiol (EE). A total of 3 patches will be worn during the study. Each patch will be worn for 1 week followed by a patch free week.
Arm/Group | AG200-15
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Steady-State Concentration (Css) (48-168) Profile for LNG
Description: Pharmacokinetic (PK) sampling will be done after exposure to each anatomic location. PK evaluations were performed at the following time points: hour (immediately prior to dosing) and at 3 hours, 6 hours, 12 hours, 24 hours (1 day), 48 hours (2 days), 72 hours (3 days), 120 hours (5 days), 144 hours (6 days), and 168 hours (7 days) following application of the patch.
Time Frame: 6 weeks
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- AG200-15: Subjects will be randomly assigned to one of six treatment (site of application) sequences. Each sequence will include three patch application sites: abdomen, buttock, or upper torso excluding breasts.
  AG200-15: A transdermal contraceptive delivery system for LNG and EE. A total of 3 patches will be worn during the study. Each patch will be worn for 1 week followed by a patch free week.
Arm/Group | AG200-15
Number analyzed (Participants) | 22
pg/mL
  Abdomen | 1256 (998)
  Buttock | 1246 (725)
  Upper torso | 1384 (728)

2. Primary Outcome: Steady-State Concentration (Css) (48-168) Profile for EE
Description: as for outcome 1
Time Frame: 6 weeks
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AG200-15
Number analyzed (Participants) | 22
pg/mL
  Abdomen | 35.8 (19.9)
  Buttock | 40.7 (16.4)
  Upper torso | 42.3 (17.0)

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) (0-168) Profile for LNG
Description: as for outcome 1
Time Frame: 6 weeks
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | AG200-15
Number analyzed (Participants) | 22
ng*hr/mL
  Abdomen | 182 (135)
  Buttock | 197 (116)
  Upper torso | 206 (106)

4. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) (0-168) Profile for EE
Description: as for outcome 1
Time Frame: 6 weeks
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | AG200-15
Number analyzed (Participants) | 22
ng*hr/mL
  Abdomen | 5.8 (2.8)
  Buttock | 7.12 (2.85)
  Upper torso | 6.86 (2.53)

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- AG200-15 on Lower Abdomen; AG200-15 on Buttock; AG200-15 on Upper Torso Excluding Breast: Subjects will be randomly assigned to one of six treatment (site of application) sequences. Each sequence will include three patch application sites: abdomen, buttock, or upper torso excluding breasts.
  AG200-15: A transdermal contraceptive delivery system for LNG and EE. A total of 3 patches will be worn during the study. Each patch will be worn for 1 week followed by a patch free week.
Arm/Group | AG200-15 on Lower Abdomen | AG200-15 on Buttock | AG200-15 on Upper Torso Excluding Breast
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 19/22 | 23/23 | 21/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG200-15 on Lower Abdomen (N=22) | AG200-15 on Buttock (N=23) | AG200-15 on Upper Torso Excluding Breast (N=23)
Gastrointestinal disorders (Gastrointestinal disorders) | 6 (6) | 12 (12) | 10 (10)
General disorders and adminstration site conditions (General disorders) | 7 (7) | 7 (7) | 13 (13)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Nervous system disorders (Nervous system disorders) | 8 (8) | 11 (11) | 7 (7)
Psychiatric disorders (Psychiatric disorders) | 3 (3) | 3 (3) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 9 (9) | 13 (13) | 10 (10)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Vascular disorders (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Approval by Agile Therapeutics, Inc. of any publication, including oral presentations and abstracts, utilizing data or any information from the ATI-CL15 study is required prior to publication submission.